CLINICAL TRIAL: NCT06135246
Title: Efficacy of High-Intensity Laser Therapy in the Management of Venous Leg Ulcers: A Randomized Controlled Trial
Brief Title: Laser Therapy for Venous Leg Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Director of Electromyography lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VLU-HILT-2023
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Venous Leg Ulcer; Varicose Ulcer; Stasis Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care group (Active Comparator): Participants will receive standard compression bandaging and wound care alone without high-intensity laser therapy. Bandaging will be applied weekly and wound care will be performed as per institutional protocols.
  Interventions: Other: Standard Care
- High Intensity laser therapy + Standard care group (Experimental): Participants will receive high-intensity laser therapy 3 times per week for 8 weeks or until ulcer closure in addition to standard care.
  Interventions: Device: High Intensity Laser Therapy; Other: Standard Care

INTERVENTIONS:
Device: High Intensity Laser Therapy — Participants will receive high-intensity laser therapy using an 810nm continuous wave diode laser (Multiwave locked System (MlS) provided by aSa). The laser applicator has a flat top hat beam profile with a spot size of 1cm2. The laser will be delivered in direct contact mode perpendicularly to the ulcer surface. Each 1cm2 area of the venous ulcer and a 1cm margin of periwound skin will be treated sequentially using a overlapping grid pattern to cover the entire ulcer area, with a 1 second exposure time per point. This results in a laser energy density of 4J/cm2 delivered to each point.
  Other Names: HILT
  Arms: High Intensity laser therapy + Standard care group
Other: Standard Care — Participants will receive standard compression bandaging and wound care as per institutional protocols, without any laser therapy. The compression bandaging protocol is based on recommendations from the American Venous Forum and American College of Phlebology guidelines (O'Donnell et al., 2014). Multi-layer compression bandages will be applied weekly by trained nurses, with layers including orthopedic padding, elastic bandages, and cohesive bandages. Bandages will be applied with high pressure at the ankle gradually decreasing up the leg, with an ankle pressure of approximately 40 mmHg (Mosti et al., 2015).

SUMMARY:
This randomized controlled trial will evaluate the effects of high-intensity laser therapy on wound healing in patients with venous leg ulcers. Participants will be randomly assigned to receive either laser therapy plus standard care or standard care alone. The laser therapy will be administered 3 times per week for 8 weeks or until ulcer closure. The primary outcome is proportion of participants with complete ulcer closure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years up to 65 years.
2. Presence of a venous leg ulcer, confirmed by clinical examination and Doppler ultrasound (venous reflux > 0.5 seconds).
3. Ulcer size between 1 cm² and 20 cm² at screening.
4. Ulcer duration of at least 4 weeks but not more than 12 months.
5. Ankle-brachial index (ABI) ≥ 0.8, assessed by Doppler ultrasound.
6. Willing and able to provide informed consent and comply with study procedures.

Exclusion Criteria:

1. Presence of an active infection in the ulcer, confirmed by clinical signs and positive culture results.
2. Osteomyelitis, diagnosed by radiographs or magnetic resonance imaging (MRI).
3. Patients with a history of uncontrolled diabetes, defined as HbA1c level > 10%.
4. Current or planned use of systemic immunosuppressive drugs or corticosteroids during the study period.
5. Pregnant or breastfeeding women.
6. Patients with a history of malignancy or photosensitive skin disorders.
7. Prior history of skin grafting or flap surgery in the affected area within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-16 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in ulcer area from baseline to end of treatment | Baseline, 4 weeks, 8 weeks and 12 weeks after randomization
  Ulcer area will be measured by tracing the wound perimeter on acetate paper and entering into image analysis software to calculate area in cm2. Percent change in ulcer area will be calculated as (area at end of treatment - area at baseline) / area at baseline x 100.

SECONDARY OUTCOMES:
Rate of complete ulcer closure at end of treatment | Single time point at end of study at 12 weeks
  Complete closure is defined as full re-epithelialization of the ulcer with no drainage. Assessed by clinical examination and tracing wound area as 0cm2. Reported as proportion of participants with complete closure.
Time to complete ulcer closure | From baseline (week 0) until complete closure, up to 12 weeks.
  Number of days from initial treatment until first point at which complete ulcer closure is achieved and maintained through end of treatment period.
Changes in Quality of life | Change in total score on the Cardiff Wound Impact Schedule will be assessed from baseline (week 0), 4 weeks, 8 weeks and 12 weeks after randomization
  The Cardiff Wound Impact Schedule is a condition-specific quality of life questionnaire designed for patients with chronic wounds. It contains 15 questions assessing physical symptoms and daily living. Each item is rated on a 4-point Likert scale from 1 (never) to 4 (all the time). Total score ranges from 15 to 60, with higher scores indicating poorer quality of life.
Incidence of treatment-related adverse events | From initial treatment until 4 weeks after final treatment, up to 12 weeks total.
  Adverse events will be graded per CTCAE v4.0. Number of participants experiencing each severity grade of adverse event related to study treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.D, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided